CLINICAL TRIAL: NCT06956898
Title: The Effect of Mindfulness-Based Intervention and Haptonomy Application on Birth Self-Efficacy, Prenatal Attachment and Anxiety Levels of Pregnant Women With Fear of ChildBirth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Responsible Party: Principal Investigator, Hafsa Kübra, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14219
Record Dates: First submitted 2025-01-14; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Fear of Childbirth; Haptonomy; Mindfulness; Self-Efficacy; Attachment
Keywords: Attachment; Self-Efficacy; Mindfulness; Haptonomy; Fear of Childbirth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness Group (Experimental): Providing mindfulness training
  Interventions: Other: Mindfulness Training
- Haptonomy Group (Experimental): Providing haptonomy training
  Interventions: Other: Haptonomy Training
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Mindfulness Training — Primiparous pregnant women in the experimental (mindfulness) group will be given training for 8 weeks starting from the 28th week.
  Arms: Mindfulness Group
Other: Haptonomy Training — Primiparous pregnant women in the experimental (mindfulness) group will be given training for 8 weeks starting from the 28th week.
  Arms: Haptonomy Group

SUMMARY:
Fear of childbirth is a common condition encountered during pregnancy. Women with fear of childbirth have reduced birth self-efficacy, and it leads to mental health problems in the prenatal and postnatal periods, reducing mother-infant bonding. Therefore, it is of critical importance to implement effective and applicable interventions focused on health and well-being to reduce fear of childbirth. Considering the increasing cesarean section rates today, holistic intervention strategies that can positively affect the birth experiences of pregnant women and support their psychological well-being are needed. In this sense, mindfulness and haptonomy applications, which are holistic intervention strategies, will allow us to meet the psychological and emotional needs of pregnant women with fear of childbirth and improve their birth experiences.

No study has been found in the literature that systematically evaluates the effects of a holistic intervention strategy for women with fear of childbirth during pregnancy. This study will enable the development of new and effective intervention strategies that can be used in prenatal and postnatal care practices and will guide clinical practices to make pregnant women's birth experiences more positive. In this study, the effects of mindfulness-based intervention and haptonomy application on childbirth self-efficacy, prenatal attachment and anxiety levels in pregnant women experiencing fear of childbirth will be evaluated. This research will be conducted as a randomized controlled experimental study. The data of the research will consist of 225 women (75 in the mindfulness group, 75 in the haptonomy group, and 75 in the control group) who applied to the Erzurum City Hospital Gynecology and Obstetrics Clinic between 01.06.2024 and 01.07.2025. The data will be collected face to face using the "Personal Information Form", "Wijma Childbirth Expectation/Experience Scale Version A", "Prenatal Attachment Inventory", and "State Anxiety Scale".

ELIGIBILITY:
Inclusion Criteria:

* Being a primary school graduate,
* Women in their 28th week of pregnancy,
* Being primigravida,
* Women with a healthy pregnancy,
* Women with a Wijma Childbirth Expectation/Experience Scale version A score of ≥38,
* Women who agree to participate in the study and do not have any chronic health problems that would prevent them from participating.

Exclusion Criteria:

* Pregnant women who did not agree to participate in the study or who left the study at any stage of the study will constitute the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women will be included in the study.
Enrollment: 225 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Childbirth Fear | "Baseline (28th week of pregnancy)" and "Post-test immediately after the training" and "Post-test 2 weeks after the training"
  Change in Fear of Childbirth Measure: Wijma Delivery Expectancy/Experience Questionnaire Version A (W-DEQ-A) Description: The W-DEQ-A is a 33-item Likert-type scale developed to assess fear of childbirth, labor-related thoughts and emotions, and anticipated stress. Each item is scored from 0 ("completely") to 5 ("not at all"), with some items reverse-coded. Total scores range from 0 to 165. Higher scores indicate greater fear of childbirth.
  Unit of Measure: Score on W-DEQ-A (0-165) Time Frame: Baseline (Week 28), immediately after training (Week 37), and two weeks after training (Week 39)
Change in Childbirth Self-Efficacy | "Baseline (28th week of pregnancy)" and "Post-test immediately after the training" and "Post-test 2 weeks after the training"
  Measure: Childbirth Self-Efficacy Inventory (CSEI)
  Description: The CSEI measures women's confidence in coping with labor. It consists of 32 items divided into two subscales: outcome expectancy and efficacy expectancy. Each item is rated on a scale from 1 to 10. Total scores range from 32 to 320. Higher scores reflect greater self-efficacy during childbirth.
  Unit of Measure: Score on CSEI (32-320)
  Time Frame: Baseline (Week 28), immediately after training (Week 37), and two weeks after training (Week 39)
Change in Prenatal Attachment | "Baseline (28th week of pregnancy)" and "Post-test immediately after the training" and "Post-test 2 weeks after the training"
  Measure: Prenatal Attachment Inventory (PAI)
  Description: The PAI is a 21-item instrument used to assess a pregnant woman's emotional attachment to her unborn baby. Items are scored from 1 to 4. Total scores range from 21 to 84. Higher scores indicate stronger prenatal attachment.
  Unit of Measure: Score on PAI (21-84)
  Time Frame: Baseline (Week 28), immediately after training (Week 37), and two weeks after training (Week 39)
Change in Trait Anxiety | "Baseline (28th week of pregnancy)" and "Post-test immediately after the training" and "Post-test 2 weeks after the training"
  Measure: State-Trait Anxiety Inventory - Trait Form (STAI-T)
  Description: The STAI-T measures an individual's general tendency to experience anxiety. The scale consists of 20 items rated on a 4-point Likert scale. Total scores range from 20 to 80. Higher scores indicate higher levels of trait anxiety.
  Unit of Measure: Score on STAI-T (20-80)
  Time Frame: Baseline (Week 28), immediately after training (Week 37), and two weeks after training (Week 39)

OTHER OUTCOMES:
Personal Information Form | "Baseline (28th week of pregnancy)"
  This form was developed by the researchers based on the relevant literature. It is used to collect the socio-demographic and obstetric information of the participants and their perceptions about birth. Data obtained will be used to describe sample characteristics and for subgroup analysis purposes. It is not considered a primary or secondary outcome measure.
  The topics covered are; Age group, Educational status, Employment status, Income level, Last menstrual period, Week of gestation, Whether the pregnancy was planned or not, Access to prenatal care, Labor pain and fear of childbirth, Attitudes towards awareness, haptonomy and perceived effectiveness of prenatal care in reducing fear of childbirth
  Participants respond using multiple choice or yes/no options. Responses will be analyzed descriptively and used to investigate associations with primary outcomes where appropriate.
  Baseline (28th week of pregnancy)

IPD SHARING:
Plan to Share IPD: No
The research is still in the implementation phase.